CLINICAL TRIAL: NCT01040338
Title: Functional Characterization of OPRM1 A118G in Nicotine Dependence: IV Nicotine Study
Brief Title: Effects of Nicotine on Brain Opioid Receptors
Status: Terminated | Type: Observational
Why Stopped: Issues & unreliability with [11C]Carfentanil production
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 809187; R21DA027066 (NIH)
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Nicotine Dependence
Keywords: Smoking; Tobacco; Nicotine; Dependence; Genetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Nicotine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples that shall be collected for this study are as follows:
  1. A 2ml saliva sample will be collected for DNA extraction using the Oragene™ kit at the Medical screening session for genetic analyses.
  2. An additional saliva sample (~ 5ml) will be also be collected at Medical screening and will be used to analyze baseline nicotine metabolites (i.e., cotinine and 3-hydroxycotinine).
  3. All participants will provide two tubes of blood (10 ml each) to measure plasma estradiol & cortisol levels before each PET scanning session. They will also provide two tubes of blood (10 ml each) at the end of the scan to measure plasma nicotine and cortisol levels.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- OPRM1 A118G AA genotype: Individuals with the AA genotype at the OPRM1 A118G polymorphism.
  Interventions: Drug: Nicotine
- OPRM1 A118G AG or GG genotype: Individuals with the */G allele at the OPRM1 A118G polymorphism
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Participants shall receive an intravenous injection of nicotine during their practice session and one of their PET scans (double-blind). The dose of IV nicotine will be 1mg/70kg and the maximum dose that shall be injected is 1.2mg.

SUMMARY:
A substantial body of evidence implicates the endogenous opioid system, and the mu opioid receptor (MOR) in particular, in the reinforcing effects of drugs of abuse, including nicotine. A single nucleotide polymorphism (SNP) in the mu opioid receptor gene (OPRM1 Asp40) is associated with the ability to quit smoking, as well as nicotine reward and withdrawal symptoms. However, the precise mechanism through which this SNP influences nicotine dependence remains unresolved. This positron emission tomography (PET) study will examine whether this OPRM1 SNP alters MOR binding in response to nicotine in human smokers. Specifically, we will use [11 C]carfentanil PET imaging to assess the effects of intravenous (IV) nicotine versus saline (within-subject) on MOR binding potential in 24 chronic smokers genotyped prospectively and stratified by OPRM1 genotype.

DETAILED DESCRIPTION:
The study uses a mixed factorial design with one between subject factor (OPRM1 genotype_: Asn40/Asn40 vs. Asn40/Asp40 or Asp40/Asp40) and one within-subject factor (IV nicotine vs. IV saline) to examine genotype by nicotine interactions on MOR binding potential (BP_ND ) assessed via PET imaging with [11 C]carfentanil. Twenty-four smokers (12 male, 12 female; 12 from each genotype group) will participate in two 90 minute PET sessions following overnight (14-hours) abstinence from nicotine. Genotype groups will be matched for age and sex . One week prior to the first PET session, there will be an adaptation session during which participants will receive IV saline followed 30 minutes later by IV nicotine (1 mg/70 kg) to ensure that they tolerate the procedure. In the PET sessions, participants will receive either IV nicotine (1 mg/70 kg) or saline (within-subject, double blind, counterbalanced). The primary outcomes will be BP_ND in ventral striatum and anterior cingulate cortex (ACC). Normally menstruating women will be scheduled for their sessions during the early follicular phase. Sessions will be separated by 1 month for all participants to reduce variability in MOR binding due to hormonal changes during females menstrual cycles. Participants will complete subjective measures of nicotine reward and craving at each session.

ELIGIBILITY:
Inclusion Criteria:

* Non-treatment seeking smokers of European ancestry
* Between 18 and 50 years old
* Smoking at least 10 cigarettes per day for at least the past 6 months
* Able to provide informed consent
* Fluent, English-speaking
* Weight ≤ 300 lbs.

Exclusion Criteria:

* Current enrollment or plans to enroll in a smoking cessation program, or use other smoking cessation medications in the next 2 months
* Provide a Carbon Monoxide reading of ≤10 ppm at Medical screening.
* History of substance abuse and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, or stimulants)
* Current alcohol consumption that exceeds 25 standard drinks/week
* Providing a breath alcohol concentration (BAC) reading of > 0.01 at any session.
* Women who are pregnant, planning a pregnancy, or lactating; all female subjects shall undergo a urine pregnancy test at each session
* Women of child-bearing age must agree in writing to use an approved method of contraception
* History or current diagnosis of psychosis, major current depression or bipolar disorder, ADHD, schizophrenia, or any Axis 1 disorder as identified by the MINI
* Serious or unstable disease within the past 6 months (e.g., cancer [except melanoma], heart disease, HIV)
* History of epilepsy or a seizure disorder
* History or current diagnosis (last 6-months) of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of COPD, cardiovascular disease (stroke, angina, coronary heart disease), heart attack in the last 6 months, uncontrolled hypertension (SBP>150 or DBP>90)
* Any medical or neurological condition that might interfere with the distribution of the radiotracer as determined by the study MD
* Current or past use (within past 12 months) of any medications containing naltrexone or other MOR antagonists (e.g., Revia, Trexan)
* Current use or recent discontinuation (within last 14-days) of the following medications
* Any form of smoking cessation medication (Zyban, Wellbutrin, Wellbutrin SR, Chantix, NRT)
* Recent (within last 2 weeks) or planned use of psychotropic medications (anti-psychotics, anti-depressants (tricyclic, SSRI, MAOI), anti-anxiety or panic medications, and stimulants (e.g., Provigil, Ritalin), and opiate-containing medications for chronic pain
* Allergic response to any form of opioids or naloxone
* Participants shall be instructed to refrain from using any study prohibited drugs (note - participants are allowed to take prescription medicines not in the exclusion list) throughout their participation in the study.
* Self-reported history of head trauma or prior seizure, brain (or CNS) tumor
* Self-reported history of claustrophobia (contraindicated for PET)
* Inability to complete the baseline study procedures within four hours and/or correctly, as determined by the principal investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 adult, non-treatment seeking smokers of European ancestry, reporting consumption of ≥10 cigarettes per day for at least the past 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
MOR binding potential | 5/31/2011

SECONDARY OUTCOMES:
Subjective reward/liking and cravings to smoke | 5/31/2011

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Center website — http://www.med.upenn.edu/tturc/